CLINICAL TRIAL: NCT03667066
Title: Prevalence of clOpidogrel "resIstaNce" in a Selected Population of Patients Undergoing Elective Percutaneous Coronary Intervention at a Tertiary Cardiovascular Center in Trinidad: The POINT Pilot Study
Brief Title: clOpidogrel "resIstaNce" in a Selected Population of Patients at a Tertiary Cardiovascular Center in Trinidad
Acronym: POINT
Status: Completed | Type: Observational
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Other Study IDs: CEC057/11/15
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Platelet Dysfunction
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Clopidogrel — Patients who were on long-term (more than 3 months) of clopidogrel or received a loading dose more than 4 hours prior to elective percutaneous coronary intervention.

SUMMARY:
The aim of this study was to determine the prevalence of clopidogrel resistance among a selected group of patients undergoing elective percutaneous coronary intervention and to observe whether there was any south-Asian (Indo-Trinidadian) predilection for HPR considering the well-established epidemiologic trends for accelerated CAD within this subgroup.

DETAILED DESCRIPTION:
Clopidogrel, a second generation oral thienopyridine, remains an integral component of dual antiplatelet therapy (DAPT) in the management of cardiovascular disease (CVD) for almost two decades. Several studies underscore the importance of high on-treatment platelet reactivity (HPR) as a prognosticator for cardiovascular events including stent thrombosis. This phenomenon is often alluded to as "clopidogrel resistance" and yet to be clearly defined. Generally, it reflects the failure to achieve its antiaggregatory effect. Clopidogrel response is both complex and multifactorial, determined by a multitude of intrinsic and extrinsic mechanisms including genetic polymorphisms of the P2Y12 receptor, drug-drug interactions, and clinical factors such as suboptimal dosing regimens, acute coronary syndromes, diabetes mellitus, and possibly smoking.

High pre-treatment platelet reactivity may lead to mitigated clopidogrel-induced antiplatelet effects and are more commonly observed in specific clinical scenarios such as ACS, increased body mass index, and diabetes mellitus, in particular, insulin-dependent diabetes mellitus. Matetzky et al also surmised that nearly one-quarter of ST-segment elevation acute coronary syndrome patients would incur stent thrombosis due to this phenomenon.

Overall, HPR prevalence in various studies is estimated at 5%-44%, however, these are based on largely Caucasian populations and yet to be ascertained in a Caribbean subpopulation. Trinidad and Tobago has an ethnically diverse population with approximately one-third South Asian (Indo-Trinidadian), one-third Caribbean Black (Afro-Trinidadian) and the remaining one-third, mostly interracial and mixed. CVD is currently the leading cause of mortality in Trinidad and Tobago, accounting for up to 60% of all deaths annually.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* diagnosed with stable angina awaiting elective coronary angiography on dual antiplatelet therapy for at least 3 months with aspirin 81 mg per day maintenance dose and "brand name" clopidogrel 75 mg per day maintenance dose

Exclusion Criteria:

* generic clopidogrel, i.e. not "brand name,"
* recent acute coronary syndrome within 6 months
* active bleeding
* prior cerebrovascular event
* clinical instability after an index event
* use of an oral anticoagulation agent (coumadin derivative or other anticoagulant therapy (such as dabigatran, rivaroxaban or apixaban)
* platelet count < 100 x 106/µL
* hemoglobin < 10 g/dL
* serum creatinine > 2.5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional, open-label (Plavix, Sanofi SA, Gentilly, France, Bristol-Myers Squibb, New York, USA) pilot study aimed to assess high on-treatment platelet reactivity which occurred during the period September 2017 to January 2018. Patients were screened with a stratified permuted block randomization technique which applied to both recruitment days (Monday, Tuesday and Thursday) and patients enrolled at the cardiac catheterization laboratory (cardiac bays 1 to 4) at the investigator's institution (Eric Williams Medical Sciences Complex, Trinidad and Tobago). The clinical research associates were blinded to the allocation assignment and randomization sequence numbers were obtained from SPSS version 24.0 software (IBM SPSS Statistics, New York City, New York, USA). On average, 1-2 patients were enrolled every week for 8 months.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Overall prevalence of HPR in the Trinidadian population undergoing elective percutaneous coronary intervention | 4 months

SECONDARY OUTCOMES:
Prevalence of HPR in the South Asian Trinidadian population undergoing elective percutaneous coronary intervention | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Naveen A Seecheran, MBBS MSc, Principal Investigator — The University of The West Indies
Locations (1):
- Eric Williams Medical Sciences Complex, Port of Spain, North, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: Yes
All information will be shared with requesting parties.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It will be openly available until 5 years after the completion of the study.
Access Criteria: Please contact the Principal Investigator for the requested information.

REFERENCES:
- [Derived] Seecheran NA, Maharaj A, Boodhai B, Seecheran R, Seecheran V, Persad S, Ramsaroop K, Sandy S, Giddings S, Sakhamuri S, Ali R, Motilal S, Teelucksingh S, Tello-Montoliu A. Prevalence of clOpidogrel 'resIstaNce' in a selected population of patients undergoing elective percutaneous coronary intervention at a tertiary cardiovascular centre in Trinidad: the POINT pilot study. Open Heart. 2019 Feb 27;6(1):e000841. doi: 10.1136/openhrt-2018-000841. eCollection 2019. PMID 30997117